CLINICAL TRIAL: NCT02715492
Title: Role of (LMWH) in Prevention of Thromboembolic Complication After (TACE) in Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, MD liver diseases, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LMWH TACE
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: HCC
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarterial Chemoembolization (Active Comparator): 1st group: included 20 patients with HCC treated by TACE only.
  Interventions: Procedure: TACE
- TACE and LMWH (Experimental): 2nd group: included 20 patients with HCC treated by TACE and adjuvant dose of Low Molecular Weight Heparins (LMWH).
  Interventions: Drug: LMWH; Procedure: TACE

INTERVENTIONS:
Drug: LMWH — (Enoxheparin) 1 IU/kg per dose twice daily for 2 weeks from the 1st day of TACE
  Other Names: Enoxaparin
  Arms: TACE and LMWH
Procedure: TACE — Trans arterial chemoembolization

SUMMARY:
Hepatocellular carcinoma (HCC) is a major health problem worldwide, and most cases are inoperable because of late presentation and underlying cirrhosis. It represents the fifth most common tumor in the world and the third most frequent cause of mortality amongst patients with cancer.

Due to the worldwide difficulties in finding liver for transplantation, hepatic resection (HR) represents the main stay of curative treatment for patients with HCC. Transcatheter arterial chemoembolization (TACE) is widely used as alternative treatments for unresectable HCC or for patients not eligible to be operated on .

TACE also could be an adjuvant therapy for resectable HCC patients after hepatectomy, which could prevent recurrence and improve long-term survival .

DETAILED DESCRIPTION:
Thromboembolism is a well-recognised complication of malignant disease. Clinical manifestations vary from venous thromboembolism to disseminated intravascular coagulation and arterial embolism. Disseminated intravascular coagulation is most commonly observed in patients with haematological malignant disorders and those with wide spread metastatic cancer, whereas arterial embolism is most commonly observed in patients undergoing chemotherapy and in those with non-bacterial thrombotic endocarditis .

The goals of using antithrombotic therapy with TACE in HCC are to minimize mortality and to improve survival rate without provoking excessive bleeding.

ELIGIBILITY:
Inclusion Criteria:

* HCC which was not amenable to surgical resection, liver transplantation or local ablative therapy.
* The lesion had not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* Reasonable performance status as adequate hematologic function; adequate hepatic function and adequate renal function.
* Child-Pugh class A or B and no portal vein thrombosis.

Exclusion Criteria:

* Child C patients Portal vein thrombosis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with portal vein thrombosis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Osama Negm, Prof, Principal Investigator — Prof. liver diseases-Tanta university; Sabry Abou Saif, Ass. Prof., Study Chair — Ass/ Prof. liver diseases-Tanta university; Mohamed El Gharib, Ass. Prof., Study Director — Ass. Prof. interventional radiology - Ain-shams university; Sherief Abd-Elsalam, Lecturer, Study Director — MD liver diseases - Tanta university
Locations (1):
- Tanta university - faculty of medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No